CLINICAL TRIAL: NCT05658029
Title: An Investigator-initiated Study to Evaluate Safety and Efficacy of ARINA-1 in Patients With a Tracheostomy
Brief Title: An Investigator-initiated Study to Evaluate Safety and Efficacy of ARINA-1 in People With a Tracheostomy
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated due to enrollment challenges
Sponsor: Matthew Bruehl (Other)
Collaborators: Renovion, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Matthew Bruehl, M.D., WakeMed Health and Hospitals
Organization: WakeMed Health and Hospitals (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WMD-001
Record Dates: First submitted 2022-11-30; First posted 2022-12-20 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Tracheostomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open label treatment group (Experimental)
  Interventions: Drug: ARINA-1

INTERVENTIONS:
Drug: ARINA-1 — Fixed-dose solution of ascorbic acid and reduced glutathione nebulized twice daily for 4 weeks (28 days)

SUMMARY:
The goal of this investigator-initiated, open label study is to evaluate the safety and efficacy of ARINA-1 in people with a tracheostomy.

Participants will attend study visits at Screening, Baseline, Day 14, Day 28, and Day 56. There will be 3 safety phone calls at Days 2, 7, and 21. Participants will nebulize the ARINA-1 solution twice daily for 28 days

ELIGIBILITY:
Inclusion Criteria:

1. Tracheostomy for ≥6 months with no anticipated changes to tracheostomy status within the next 3 months from screening visit
2. Males or females 18-75 years old at time of consent
3. Willing and able to comply with the protocol and visit schedule
4. Subject or legal authorized representative capable of giving informed consent. Determination of subject capacity to give informed consent will be determined by investigators and guided by principles set forth in the Declaration of Helsinki (World Medical Association, 2013) and by WakeMed Health & Hospitals guidance (Patient Competency and Decisional Capacity - Legal Affairs Tip Sheet/FAQ).

Exclusion Criteria:

1. Inability to speak or understand English
2. Positive urine pregnancy test at screening and/or baseline visit, if applicable
3. Active breastfeeding status
4. Diagnosis of cystic fibrosis or primary ciliary dyskinesia
5. History of lung transplant
6. Listed for lung transplant
7. Inability to tolerate nebulized treatments
8. Planned decannulation before completion of this study
9. Exacerbation or infections requiring any acute antibiotics, urgent care visit, emergency department visit or hospitalization within 14 days of screening visit
10. Previous intolerance to hypertonic saline (HTS)
11. Initiating a chronic azithromycin or any new inhaled maintenance therapy < 28 days prior to baseline visit
12. Initiating any N-acetyl-cysteine-containing (NAC), ascorbic acid or glutathione (GSH)-containing therapy (oral or nebulized) < 28 days prior to baseline visit
13. Intolerance to NAC or GSH
14. Intolerance to bronchodilator (e.g., Albuterol)
15. Significant comorbidities that in the opinion of the investigator would reduce the safety of the subject or interfere with the ability to interpret study data
16. Currently participating in or have participated in other interventional (drug or device) clinical study within 90 days of the baseline visit
17. Receiving a vaccination within 14 days of the baseline visit

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-05-23 (Actual); Primary Completion 2023-09-09 (Actual); Study Completion 2023-09-09 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events / serious adverse events | Baseline to day 28

SECONDARY OUTCOMES:
Change from baseline to day 28 for Composite Tracheostomy Questionnaire and the Clinical Global Impression of Change (CGI-C) | Baseline to day 28
Change in mucus rheology | Baseline to day 28
Change in bacterial culture at 28 days | Baseline to day 28
Changes in blood CRP over 28 days | Baseline to day 28
Ventilator settings / respiratory system compliance (for subjects on intermittent chronic ventilatory support) | Baseline to day 28
Peripheral Oxygen Saturation (SpO2) | Baseline to day 28

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Bruehl, MD, Principal Investigator — WakeMed Health & Hospitals
Locations (1):
- WakeMed Health & Hospitals, Raleigh, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No